CLINICAL TRIAL: NCT03861676
Title: Image-guided Focal Brachytherapy Utilizing Combined 18F-DCFPyl PET/CT and Dynamic Dosimetry With Registered Ultrasound and Fluoroscopy for Localized Prostate Cancer
Brief Title: Image-guided Focal Brachytherapy Utilizing Combined 18F-DCFPyl PET/CT
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J1889; IRB00173561 (Other: JHM IRB); R01CA151395 (NIH)
Record Dates: First submitted 2019-03-01; First posted 2019-03-04 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Prostate Cancer
Keywords: focal therapy; brachytherapy; PSMA; DCF-Pyl
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy; Radiation; 2-(3-(1-carboxy-5-((6-fluoropyridine-3-carbonyl)amino)pentyl)ureido)pentanedioic acid; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

STUDY DESIGN:
Intervention Model Description: Single-arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Focal brachytherapy (Experimental): Drug: 18F-DCFPyl Other names: PET, PSMA
  Procedure: Focal brachytherapy with PSMA PET imaging Other names: Radiotherapy, Radiation, Prostate seed implant, Focal therapy
  Interventions: Radiation: Focal brachytherapy with PSMA PET imaging; Drug: (18F)DCFPyL

INTERVENTIONS:
Radiation: Focal brachytherapy with PSMA PET imaging — Focal brachytherapy with PSMA PET imaging. Focal (partial prostate gland) brachytherapy following 18F-DCFPyl PET/CT radiotracer imaging. Patients will also undergo pre-treatment transperineal mapping biopsy.
  Other Names: Prostate seed implant; Radiotherapy; Radiation; Focal therapy
Drug: (18F)DCFPyL — 18F-DCFPyl PET/CT scan
  Other Names: PSMA, PET

SUMMARY:
The Principal Investigator's (PI) working hypothesis is that the PI can utilize the high predictive value of 18F-DCFPyl PSMA to identify clinically significant tumors in patients who will undergo brachytherapy, as well as areas which are uninvolved or contain only clinically insignificant disease.

In the PI's clinical trial, the uninvolved regions (as defined by combined PET-MR-biopsy data) will not be targeted and receive only fall-off dose, which we have shown to be associated with reductions in toxicity.

DETAILED DESCRIPTION:
Current conventional prostate cancer (PCa) imaging modalities (computed tomography, bone scan, magnetic resonance imaging, ultrasound) have limited accuracy in the initial staging and for determining prognosis of PCa. Prostate-specific membrane antigen (PSMA) is a cell surface antigen which is highly expressed in PCa and correlates with prognostic factors such as Gleason score. High PSMA expression in prostate tumor has been significantly associated with lethality of disease, allowing specific identification of tumors most in need of treatment. Combined PET and computed tomography (PET-CT) imaging using small molecules targeting PSMA-expressing cells have been developed and tested clinically, and have shown superiority when compared with conventional imaging.

An added advantage of PET compared to MRI is the ability to identify both distant metastatic disease as well as intraprostatic disease with one imaging modality. PSMA-radiotracers have continued to evolve since their initial development, with successive improvements in imaging and diagnostic characteristics. One such second-generation PSMA-binding compound, 18F-DCFPyl, has been developed and characterized at our institution, and offers superior imaging qualities compared to prior PSMA-based radiotracers.

In realization of the toxicity of current therapies, there is substantial interest throughout the urologic oncology community in utilizing focal therapy to mitigate such toxicities. The rationale for focal therapy is based upon the recognition that whole gland treatment is associated with unacceptable toxicity rates, while concurrently it is also realized that patient morbidity and mortality is due to the progression of major foci of high-grade disease, i.e. the index lesion.

Planning studies have shown that focal brachytherapy is feasible and results in significant reductions of dose to critical structures. In a historic cohort of patients treated at Johns Hopkins, the investigators have demonstrated that a modest reduction in dose results in clinically meaningful reductions in urinary toxicity. Al-Qaiseh et al. found that focal plans resulted in >50% reductions in dose to urethra and rectum. However, focal plans were highly sensitive to seed positioning errors, and focal targeting made seed positioning more critical. This highlights the key utility and importance of the investigators' iRUF system (integrated Registered Fluoroscopy and Ultrasound) in delivering focal therapy.

The investigators have developed a system of true dynamic intraoperative dosimetry which utilizes fluoroscopy for seed cloud reconstruction and fusion to transrectal ultrasound imaging. The investigators previously confirmed this method in a pilot trial of 6 patients with encouraging results. Further refinement of the system was followed by a Phase II clinical trial of this integrated platform on a larger group of patients. The investigators confirmed the primary endpoint to compare intraoperative dosimetric predicted values using iRUF method vs standard ultrasound-based seed tracking. The iRUF Phase II cohort had statistically significant improvements in prostate coverage parameters, as well as lower rates of rectal doses exceeding prescribed tolerance limits when compared to a historical group of patients. Importantly, there was no trend toward higher prostate V200 doses, indicating that excellent coverage did not come at the expense of excessive dose within prostate.

This study will test the combination of PSMA-imaging with iRUF dynamic dosimetry to treat prostate cancer with a focal approach.

ELIGIBILITY:
Inclusion Criteria:

* Adenocarcinoma of the prostate
* Performance Status < 2
* Clinical stages (not radiographic stage) T1c - T2a, Nx or N0, Mx or M0
* Gleason 6-7 cancer
* Prostate volume < 60 cc (if MRI and TRUS have conflicting values, then MRI value will be utilized)
* International Prostate symptom score (IPSS) 20 or less
* Ability to undergo DCF-Pyl PSMA PET as part of pretreatment staging
* Signed study-specific consent form prior to registration

Exclusion Criteria:

* Prior history of pelvic radiation therapy
* Major medical or psychiatric illness which, in the investigator's opinion, would prevent completion of treatment and would interfere with follow up.
* Implanted device or apparatus which obstruct visibility of the implanted sources on fluoroscopy
* Metallic implants, claustrophobia not amenable to medication, or known contraindications to undergoing MR scanning
* History of other malignancy diagnosed within the past 3 years

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2023-08-03 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
Percent tumor coverage | Post-implant Day 30
  Percent coverage of the combined PET-MR based tumor volume achieved when using iRUF intraoperative dosimetry.
  PET-MR tumor volume D90 will be defined on pre-treatment PET-MR fusion, and dose from seeds will be calculated on post-implant MR/CT (Day ~30); the two volumes will be co-registered to determine tumor volume coverage.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Song, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- SKCCC at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No